CLINICAL TRIAL: NCT06281704
Title: A Phase Ib Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of Single and Multiple Administration of AK101 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of AK101 in Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK101-102
Record Dates: First submitted 2021-11-25; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis
Keywords: AK101; safety; pharmacokinetics; efficacy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1 : AK101 IV (Experimental): Subjects will be enrolled in sequential cohorts treated with successively higher doses of AK101 via intravenous injection on Day1.
  Interventions: Biological: AK101 IV
- Part 1 : AK101 SC (Experimental): Subjects will be enrolled in sequential cohorts treated with successively higher doses of AK101 via subcutaneous injection on Day1.
  Interventions: Biological: AK101 SC
- Part 1 :Placebo (Placebo Comparator): Subjects will be received matching placebo intravenously or subcutaneously on Day1.
  Interventions: Biological: Placebo
- Part 2:AK101-AK101 low-dose SC every 8 weeks (Experimental): Subjects received single IV infusion of AK101 on Day1 will be randomized to receive low-dose AK101 subcutaneously every 8 weeks along with matching placebo subcutaneously (to maintain the blind).
  Interventions: Biological: AK101 SC
- Part 2: AK101-AK101 high-dose SC every 8 weeks (Experimental): Subjects received single IV infusion of AK101 on Day1 will be randomized at Week8 to receive high-dose AK101 subcutaneously every 8 weeks.
  Interventions: Biological: AK101 SC
- Part 2: Placebo-AK101 low-dose SC every 8 weeks (Experimental): Subjects received placebo on Day1 will receive a single IV infusion of AK101 at Week8 along with matching subcutaneous placebo (to maintain the blind). And subjects will be randomized at Week8 to receive low-dose AK101 subcutaneously every 8 weeks along with matching placebo subcutaneously (to maintain the blind).
  Interventions: Biological: AK101 IV/AK101 SC
- Part 2:Placebo-AK101 high-dose SC every 8 weeks (Experimental): Subjects received placebo on Day1 will receive a single IV infusion of AK101 at Week8 along with matching subcutaneous placebo (to maintain the blind). And subjects will be randomized at Week8 to receive high-dose AK101 subcutaneously every 8 weeks.
  Interventions: Biological: AK101 IV/AK101 SC

INTERVENTIONS:
Biological: AK101 IV — AK101 will be administered intravenously.
  Arms: Part 1 : AK101 IV
Biological: AK101 SC — AK101 will be administered subcutaneously.
  Arms: Part 1 : AK101 SC; Part 2: AK101-AK101 high-dose SC every 8 weeks; Part 2:AK101-AK101 low-dose SC every 8 weeks
Biological: Placebo — Placebo will be administered subcutaneously or intravenously.
  Arms: Part 1 :Placebo
Biological: AK101 IV/AK101 SC — AK101 will be administered as intravenous infusion at Week8, then subcutaneously every 8 weeks thereafter .
  Arms: Part 2: Placebo-AK101 low-dose SC every 8 weeks; Part 2:Placebo-AK101 high-dose SC every 8 weeks

SUMMARY:
This is a Phase Ib clinical study to evaluate the safety, tolerance, pharmacokinetics and efficacy of AK101 in subjects with moderately to severely active ulcerative colitis.

DETAILED DESCRIPTION:
This is a phase Ib, randomized, double-blind, placebo-controlled, dose-escalation, two-phase study evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of AK101 in subjects with moderately to severely active ulcerative colitis. The study consists of two parts. Part 1 is single-ascending-dose induction phase study, and Part 2 is a multiple subcutaneous maintenance therapy study followed by a single-dose induction treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) ≥ 18 and ≤ 28 kg /m2 for male or female patients aged between 18 and 65 years (including upper and lower limits).
* Confirmed diagnosis of ulcerative colitis (UC) for at least 3 months before screening, and the diagnosis of UC must be confirmed by endoscopic and histological evidence.
* Has moderately to severely active UC,defined as the adapted Mayo score (excluding PGA) of 5-9 (including upper and lower limits), Mayo endoscopic subscore ≥ 2 within 10 days before the first administrationof study drug and rectal bleeding subscore ≥ 1.
* Have evidence of ulcerative colitis extending proximal to the rectum (≥15 cm of involved colon).
* Demonstrated intolerance or inadequate response to conventional therapy and tofacitinib (not a biologic) and biologic therapies.
* For women with fertility, the serum pregnancy test must be negative during the screening period; Or women without fertility.If male and female subjects with sexual life and fertility voluntarily take contraceptive measures during the treatment and at least 6 months after the last Administration.

Key Exclusion Criteria:

* Suspected or confirmed Crohn's disease (CD), undiagnosed type of colitis.
* Suffering from severe generalized colitis.
* Previous colectomy (total or subtotal resection) with ileal pouch, Kock pouch or ileostomy for ulcerative colitis.
* Patients who have received IL-12 / 23 or IL-23 target drug treatment.
* Received Natalizumab or other drugs that regulate B cells or T cells within 12 months before randomization, such as Rituximab, Alemtuzumab, Abatacept treatment.
* Received infliximab and adalimumab 2 months before randomization, and received Vedolizumab and other biological treatments 3 months before randomization.
* Patients with active hepatitis B virus (HBV) infection or active hepatitis C virus (HCV).
* Suffering from human immunodeficiency virus (HIV) or syphilis.
* Active tuberculosis or Latent tuberculosis infection.
* Has a history of, or ongoing, chronic or recurrent infectious disease.,
* Suffering from any mental illness, or suffer from a serious or active disease, the investigators think may interfere with the subject's treatment, evaluation or compliance with the study protocol.
* Patients with malignant tumors (except skin basal cell carcinoma and cervical carcinoma in situ that have been cured and have no signs of recurrence) or lymphoproliferative diseases, and cervical diseases caused by HPV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From the time of signing the informed consent form till last follow-up visit (Up to Week 12 or Week36)
  Percentage of subjects with treatment-emergent adverse events (TEAEs) during the study.
Adverse Events | From the time of signing the informed consent form till last follow-up visit (Up to Week 12 or Week36)
  Percentage of subjects with treatment-emergent serious adverse events (SAEs) during the study.
Elimination half-life (T1/2) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of half-life (T1/2) of AK101
Mean residence time (MRT) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of mean residence time (MRT) of AK101
Area under curve (AUC) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of area under curve (AUC) of AK101
Apparent distribution volume (VD/F) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of apparent distribution volume (VD/F) of AK101
Systemic clearance (CL/F) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of systemic clearance (CL/F) of AK101
Maximum (peak) plasma concentration (Cmax) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of maximum (peak) plasma concentration (Cmax)
Time to maximum plasma concentration (Tmax) of AK101 | Baseline till last follow-up visit (Up to Week12 or Week36)
  Assessment of Time to maximum plasma concentration (Tmax)

SECONDARY OUTCOMES:
Proportion of subjects with clinical response at Week8(per Adapted Mayo Score without physician's global assessment). | At week 8
  Clinical response(per Adapted Mayo Score) was defined as a decrease from induction baseline in the adapted Mayo score by≥30 percent (%) and ≥ 2 points, with either a decrease from baseline in the rectal bleeding subscore ≥1 or a rectal bleeding subscore of 0 or 1. Adapted Mayo Score consists of 3 subscores (stool frequency, rectal bleeding and endoscopy findings), rated as 0 (normal) to 3 (severe). Total score was calculated as the sum of 3 subscores and values range from 0 to 9 scores.
Proportion of subjects with clinical response at Week8(per the Mayo score). | At week 8
  Clinical response(per the Mayo Score) was defined as a decrease from induction baseline in the Mayo score by ≥30 percent (%) and ≥ 3 points, with either a decrease from baseline in the rectal bleeding subscore ≥1 or a rectal bleeding subscore of 0 or 1. The Mayo Score consists of 4 subscores (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment), rated as 0 (normal) to 3 (severe). Total score was calculated as the sum of 4 subscores and values range from 0 to 12 scores.
Immunogenicity index | Baseline till last follow-up visit (Up to Week 12 or Week36)
  Number and percentage of subjects with detectable anti-AK101 antibody (ADA).

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guanzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjing People's Hospital, Tianjing, Tianjing